CLINICAL TRIAL: NCT06751433
Title: Evaluation of Clinical, Perceived and Instrumental Efficacy of a Scar Gel Versus Benchmark in Preventing Hypertrophic Scars and Improving Scar Appearance
Brief Title: Evaluation of Clinical, Perceived and Instrumental Efficacy of a Scar Gel in Preventing Hypertrophic Scars
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ORC-137032_EN-24-0252-01
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acceptability Study; Real-use Conditions; Safety and Efficacy; Topical Administration; Hypertrophic Scars; Keloid Scars
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Intervention Model Description: Clinical trial, double arm, double blind, randomized
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants of both sexes, 18 - 70 y (Active Comparator): Participants of both sexes, 18 - 70 y, who have recent scars.
  Interventions: Device: Scar gel comparator
- Exp.: Participants of both sexes, 18 - 70 y (Experimental): Participants of both sexes, 18 - 70 y, with recent scars
  Interventions: Device: Scar gel

INTERVENTIONS:
Device: Scar gel — Health care product (scar gel)
  Arms: Exp.: Participants of both sexes, 18 - 70 y
Device: Scar gel comparator — Health care product (Scar gel comparator)
  Arms: Participants of both sexes, 18 - 70 y

SUMMARY:
Evaluation of the safety and topical efficacy of a scar gel after 90 days of continuous use, comparing it to a benchmark for preventing hypertrophic scars and improving appearance, hydration and pigmentation.

DETAILED DESCRIPTION:
Evaluation of the safety and topical efficacy of a scar gel after 90 days of continuous use. Comparison of the efficacy of the investigational product with the benchmark product in preventing hypertrophic scars and improving scar appearance, as well as analyzing parameters such as skin hydration, pruritus, discomfort, and normalization of scar pigmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of both sexes aged between 18 and 70 years;
2. Participants with recent scars (<30 days);
3. Participants with phototypes III to VI according to the Fitzpatrick scale;
4. Agree to follow the trial procedures and attend the center on the days and times determined for evaluations;
5. Understand, agree to and sign the free and informed consent form.
6. Types of scars: cesarean section, breast implant or blunt cut injury.

Exclusion Criteria:

1. Pregnancy or risk of pregnancy;
2. History of atopic or allergic reactions to cosmetic products;
3. Participants who are using topical antibiotics or other skin products on the same area being evaluated;
4. Immunosuppression due to drugs or active diseases;
5. Decompensated endocrine diseases;
6. Relevant clinical history or current evidence of alcohol or other drug abuse;
7. Known history or suspected intolerance to products in the same category;
8. Intense sun exposure up to 15 days before the evaluation;
9. Patients who are using topical antibiotics or other skin products on the same area being evaluated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of clinical and perceived efficacy | 90 days
  Evaluate the prevention of hypertrophic scars after 90 days of continuous use of the investigational product. The dermatologist will perform assessments of the clinical parameters using the POSAS scale.

SECONDARY OUTCOMES:
Perceived efficacy | 90 days
  To compare the treatments of the benchmark product versus the investigational product in improving the appearance of scars, discomfort, skin hydration, itching and normalization of scar pigmentation, after 90 days of use, through a questionnaire on perceived efficacy.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Medcin Instituto da Pele Ltda, Osasco, São Paulo
  - MEDCIN, Osasco